CLINICAL TRIAL: NCT04751721
Title: Comparison of Oxidative Stress Parameters, Trace, Element and Quality of Life Levels in Healthy Women Before and After Covid-19 Vaccines
Brief Title: Oxidative Stress Parameters, Trace Element and Quality of Life in Women Before and After Covid-19 Vaccines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Cigli Regional Training Hospital (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021-01-173
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Covid-19 Vaccine
Keywords: Covid-19; CoronaVac vaccine; Healthy women
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoronoVac Vaccine Group (Experimental)
  Interventions: Biological: CoronoVac Vaccine

INTERVENTIONS:
Biological: CoronoVac Vaccine — CoronaVac vaccines will be inoculated in 2 doses with an interval of 24 days.

SUMMARY:
There is no effective treatment method for COVID-19 yet. With vaccination being the most effective approach to control the COVID-19 pandemic, vaccines have been developed with many different methods. One of the vaccines developed, the China-based CoronaVac vaccine (inactivated + aluminum adjuvant vaccine) is a vaccine developed with the inactive method, which is the classical vaccine production method. As a result of Phase 1, Phase 2 and Phase 3 trials, emergency use approval has been given for the CoronaVac vaccine by Turkish Pharmaceuticals and Medical Devices Agency. The clinical picture of COVID-19 can be heterogeneous, ranging from asymptomatic to severe disease, which can be associated with a cytokine storm. In the clinical results of COVID-19, it has been observed that the severity of the disease is lower in women than in men, and the mortality rates are lower in women than in men. A few studies have shown the physiological roles of some vitamins and trace elements in COVID-19. Investigation of free radical levels known to be effective in the development of cardiovascular disease due to oxidative stress is important in determining the risk of cardiovascular complications in the COVID-19 pandemic. In addition, the social isolation rules and quarantine measures applied in the COVID-19 pandemic have caused individuals to be negatively affected physically and psychologically and their quality of life to decrease. Investigating the changes in oxidative stress parameters, trace element and quality of life levels of vaccination in COVID-19 may provide useful information in determining the effects of COVID-19 vaccine. It is planned to include female individuals to be vaccinated in Izmir Bakırcay University Cigli Training and Research Hospital. Within the scope of the study, it was planned to determine the oxidative stress parameters, trace element levels and quality of life levels of the individuals and to compare the values of the data obtained before and after vaccination. After analyzing the data obtained from the research with appropriate statistical methods, the data will be evaluated.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) pandemic, also known as Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), caused by a coronavirus strain that is a member of the Betacoronavirus genus, affecting billions of people worldwide, has become a global health problem. Since vaccination is the most effective approach to control the COVID-19 pandemic, trials of many different vaccines have been started.

According to the data of the World Health Organization, there are 236 vaccines in total, with clinical (63) and pre-clinical (173) studies developed using 10 different methods.Types of vaccines for COVID-19 include conventionally live attenuated viruses, inactivated virus protein or polysaccharide conjugated subunit vaccines, virus-like particles (VLPs), nucleic acid (DNA and RNA), viral vectors (replicating and non-replicating), and the other vaccines composed of eccombinant proteins.

CoronaVac vaccine (inactivated + aluminum adjuvant vaccine) is a vaccine developed by the biopharmaceutical company named Sinovac Biotech Ltd. based in China, using the classical vaccine production method (inactive method). After the completion of Phase 1 and Phase 2 trials of the vaccine, Phase 3 trials were initiated in Turkey. Emergency use approval has been given for the CoronaVac vaccine by Turkish Pharmaceuticals and Medical Devices Agency after the end of these trials.Although the pathogenesis of COVID-19 is not fully understood, its clinical presentation may become heterogeneous, ranging from asymptomatic to severe disease.

It has been reported that a systemic hyperinflammatory response and associated thromboembolic complications are observed in cases with severe symptoms. In addition, it has been observed that the severity of the disease and mortality rates are lower in women compared to men in the clinical results of COVID-19.

The roles of vitamins A, B, C, D, E and folate and trace elements such as iron, zinc, magnesium, selenium and copper in supporting the immune system have been shown to have positive effects on COVID-19 disease.

Intermediates in enzymatic reactions occurring during cell metabolism (reactive oxygen species and reactive nitrogen) sometimes leak from the active site of enzymes and accidentally interact with molecular oxygen and form free oxygen radicals. Oxidative stress caused by free oxygen radicals forms the molecular basis in the development of cancer, neurodegenerative and cardiovascular diseases, diabetes and autoimmune disorders.

Social isolation rules and quarantine measures have negatively affected the daily lives of individuals physically and psychologically. In particular, the increase in the time spent at home causes individuals to have a sedentary life and cause their physical levels to decrease. This situation caused individuals to be psychologically affected by concerns about health, news watched, and the increasing number of cases day by day.

Studies have also reported negative psychological effects such as post-traumatic stress symptoms, confusion, disappointment, feeling of isolation and anger as a result of quarantine. These psychological and physical effects caused by the COVID-19 pandemic caused a decrease in the quality of life of individuals. During the COVID-19 pandemic, it has been reported that the depression and anxiety levels of healthcare workers increased and their quality of life decreased.

The aim of this study is to compare and determined and the changes of oxidative stress parameters, trace element and quality of life levels in healthy women just before the first dose of COVID-19 vaccine and on the 7th day after the second dose of COVID19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Agree to voluntarily participate in the study

Exclusion Criteria:

* Have been taking trace element supplements for the past 2 weeks
* Being pregnant
* Body mass index over 40 kg/m2
* Diagnosed with Covid-19 in advance
* Not diagnosed with any chronic disease

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change of the levels of Oxidative Stress Parameter 1 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameter including Superoxide Dismutase (SOD) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 2 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameters including Malondialdehyde (MDA) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 3 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameter including Total Antioxidant Level (TAL) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels of Oxidative Stress Parameter 4 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Oxidative Stress Parameters including Total Oxidant Level (TOL) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of the levels serum trace element 1 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including zinc levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 2 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace elements including selenium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 3 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including potassium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 4 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including sodium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 5 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace elements including calcium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 6 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including magnesium levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels serum trace element 7 | Immediately before the first dose and 7 days after the second dose of CoronaVac vaccine
  Serum trace element including copper levels will be determined by venous blood samples taken from the participants. Serum trace element levels samples will be analyzed using the atomic absorption spectrophotometry (AAS) method.
Change of the levels of quality of life | Immediately before the first dose and 4 weeks later
  SF-36 Quality of Life Scale will be used to determine the quality of life level. The scale that patients can apply themselves and in a short time; It consists of 36 items and 8 subsections. These sections are physical functionality, social functionality, role restrictions due to physical problems, role restrictions due to emotional problems, pain, energy level / vitality / vitality, mental health, and general health perception (40). The last 4 weeks are considered in the evaluation of the scale. The scale gives a separate total score for each subsection. The points obtained from the subsections are not added up. Subdivisions rate health from 0 to 100. While it expresses bad health status as "0 points", it refers to good health status as "100 points".

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)